CLINICAL TRIAL: NCT01550094
Title: Evaluation of Ultrasound-Guided Popliteal Sciatic Nerve Blockade in the Severely and Morbidly Obese Populations
Brief Title: A Comparison of Two Injection Locations in Obese Patients Having Lower Leg/Foot Surgery
Status: Completed | Type: Observational
Sponsor: Jose Soberon, MD (Other)
Responsible Party: Sponsor-Investigator, Jose Soberon, MD, Anesthesiologist, Ochsner Health System
Organization: Ochsner Health System (Other)
Other Study IDs: 2011.191.B; 2011.191.B (Other: Ochnser Clinic Foundation Institutional Review Board)
Record Dates: First submitted 2012-03-07; First posted 2012-03-09 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Strain of Muscle and/or Tendon of Lower Leg; Fracture of Lower Leg; Crushing Injury of Lower Leg; Fracture Malunion - Ankle and/ or Foot; Complete Tear, Ankle and/or Foot Ligament; Pathological Fracture - Ankle and/or Foot; Loose Body in Joint of Ankle and/or Foot
Keywords: obese; regional anesthesia; anesthesia; anesthesiology; surgery; foot; foot surgery; ankle; ankle surgery; orthopedics; orthopedic surgery; sports medicine; sports medicine surgery; Ochsner Hospital; Ochsner Clinic; New Orleans; Louisiana; Jefferson; Soberon
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
One technique for the nerve block involves injecting the numbing medicine where the nerve is together (higher up in the back of the thigh). The other technique involves injecting the numbing medicine where the nerve splits into two parts. By injecting numbing medication around the nerve(s), there will be less pain after the procedure. It is thought that the numbing medicine will be easier to inject in the group that the nerves are split. It is expected that subjects may need less pain medication and have lower pain ratings in this group too.

DETAILED DESCRIPTION:
The purpose of this study is to compare two different techniques for placement of nerve blocks for your foot or ankle procedure. A nerve block involves injecting numbing medications around a nerve to decrease pain after surgery. An ultrasound machine is often used to help see the nerve before injecting the numbing medicine. When an ultrasound machine is used during a block it is called an ultrasound-guided block.

Many studies of ultrasound-guided nerve blocks have involved mostly thin patients, especially from foreign countries. This study is different because the investigators are looking at patients living in America with a body mass index (a measure of the amount of body fat a person has) of more than 35.

The Sciatic nerve is a large nerve that provides most of the feeling and all of the movement to the foot and ankle. The nerve travels under the back of the leg, and splits into two smaller nerves slightly above the knee.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age undergoing unilateral foot and/or ankle surgery
* Severe or morbid obesity, defined as a BMI of 35-39 or ≥ 40, respectively
* ASA status I-IV
* Ability to understand and provide informed consent

Exclusion Criteria:

* True allergy, not sensitivity, to any of the following substances:

Local Anesthetics Midazolam Fentanyl Hydromorphone Propofol

* Pregnancy
* Evidence of infection at or near the proposed needle insertion site
* Unstable or undetermined neurologic disease of the lower extremity
* Chronic pain patients
* Patient refusal or inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Severely and morbidly obese patients scheduled for foot or ankle surgery.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2012-03; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jose Soberon, MD, Principal Investigator — Ochsner Health System
Locations (1):
- Ochsner Clinic Foundation, New Orleans, Louisiana, United States